CLINICAL TRIAL: NCT03038152
Title: A Prospective, Open Label Study of the Use of Magseed® and Sentimag® to Localize Axillary Lymph Nodes With Biopsy-Proven Metastases in Breast Cancer Patients
Brief Title: Magseed Magnetic Marker in Locating Axillary Lymph Nodes in Patients With Breast Cancer Undergoing Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0806; NCI-2017-00649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0806 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-25; First posted 2017-01-31 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Breast Carcinoma Metastatic in Lymph Node; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Magseed marker) (Experimental): Patients receive the Magseed marker via ultrasound guided injection into the previously clipped lymph node or within perinodal tissue =< 3mm from the clipped node. Patients then undergo axillary lymph node localization and targeted dissection within 30 days.
  Interventions: Procedure: Axillary Lymph Node Dissection; Procedure: Localization; Device: Medical Device

INTERVENTIONS:
Procedure: Axillary Lymph Node Dissection — Undergo targeted axillary lymph node dissection
  Other Names: ALND; Axillary Dissection; Axillary Lymphadenectomy; Axillary Node Dissection; Excision Axillary Lymph Nodes
Procedure: Localization — Undergo axillary lymph node localization
Device: Medical Device — Receive Magseed via ultrasound guided injection
  Other Names: Device; Medical Devices

SUMMARY:
This phase IV trial studies the side effects of the Magseed magnetic marker and how well it works in locating lymph nodes in the underarm area in patients with breast cancer undergoing surgery. Injecting a small metallic marker in or near the lymph node prior to surgery may help the surgeon locate the lymph nodes during surgery without using radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To provide evidence that the clipped lymph node and Magseed can be successfully retrieved in the excised surgical specimen when Magseed and Sentimag are used for targeted axillary dissection in breast cancer patients.

OUTLINE:

Patients receive the Magseed marker via ultrasound guided injection into the previously clipped lymph node or within perinodal tissue =< 3 mm from the clipped node. Patients then undergo axillary lymph node localization and targeted dissection within 30 days.

After completion of study, patients are followed up within 6-22 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cT0-4, N1 breast cancer
* Axillary lymph node metastasis with pathologic confirmation by needle biopsy
* Clip placed in the sampled axillary lymph node before completing chemotherapy
* Received neoadjuvant chemotherapy prior to surgical resection
* Scheduled for targeted axillary dissection (defined as selective localization and removal of the clipped node and sentinel lymph node dissection [SLND])
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Distant metastases
* Inflammatory breast cancer
* Prior surgical axillary procedure including SLND or axillary node excision
* Prior history of breast cancer in the ipsilateral breast
* History of lymphoma
* The subject is known to be pregnant. Premenopausal patients under the age of 50 must have a pregnancy test performed as standard of care before the MagSeed is placed
* Previous radiation to the breast or axilla
* Pacemaker of other implantable device in the chest wall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Retrieval rate | Up to 15 months
  Will be defined as the number of subjects in whom the clipped node and Magseed are retrieved in a single excised specimen divided by the total number of subjects. For the analysis of retrieval rate, if the trial is not stopped early and all 50 patients are accrued, then point estimate along with 95% credible interval will be provided. Logistic regression model will be utilized to assess the association of patient demographic and clinical factors with the retrieval.
Incidence of adverse events | Up to 6 weeks post-procedure
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Toxicity data will be summarized by frequency tables. For the toxicity endpoint, per-treated analysis will be used to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.

SECONDARY OUTCOMES:
Radiologist rated ease of Magseed placement | Up to 15 months
  Descriptive statistics will be used to summarize the radiologist rated ease of Magseed placement. Logistic regression models and/or linear regression models will be used to assess the association of variables with patient's characteristics in multivariate setting. Other statistical methods, when appropriate, may be used for analysis.
Accuracy of Magseed placement | Up to 15 months
  Will be defined as accurate, marginal or inadequate. Descriptive statistics will be used to summarize accuracy of placement. Logistic regression models and/or linear regression models will be used to assess the association of variables with patient's characteristics in multivariate setting. Other statistical methods, when appropriate, may be used for analysis.
Surgeon rated ease of node localization and removal | Up to 15 months
  Descriptive statistics will be used to summarize surgeon rated ease of localization. Logistic regression models and/or linear regression models will be used to assess the association of the above mentioned variables with patient's characteristics in multivariate setting. Other statistical methods, when appropriate, may be used for analysis.
Number of nodes retrieved within the surgical specimen containing the Magseed | Up to 15 months
  Descriptive statistics will be used to summarize number of nodes retrieved within the surgical specimen containing the Magseed. Logistic regression models and/or linear regression models will be used to assess the association of the above mentioned variables with patient's characteristics in multivariate setting. Other statistical methods, when appropriate, may be used for analysis.
Transcutaneous detection rate | Up to 15 months
  Descriptive statistics will be used to summarize transcutaneous detection rate. Logistic regression models and/or linear regression models will be used to assess the association of the above mentioned variables with patient's characteristics in multivariate setting. Other statistical methods, when appropriate, may be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail S Caudle, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org